CLINICAL TRIAL: NCT00074958
Title: A Multi-center, Phase 2, Open-Label Study of Fabrazyme (Recombinant Human a-Galactosidase A) Replacement Therapy in Pediatric Patients With Fabry Disease
Brief Title: A Study of Fabrazyme in Pediatric Patients With Fabry Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Medical Monitor, Genzyme Corporation
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGAL-016-01
Record Dates: First submitted 2003-12-24; First posted 2003-12-25 (Estimated); Results first posted 2009-06-16 (Estimated); Last update posted 2015-04-02 (Estimated); Status verified 2015-03

CONDITIONS: Fabry Disease
Keywords: a-Galactosidase A; aGal; r-haGAL; Fabry; GL-3; Fabrazyme
MeSH Terms: conditions — Fabry Disease | interventions — agalsidase beta

ARMS (1):
- Fabrazyme (Experimental): 1.0 mg/kg of Fabrazyme given to the patients every 2 weeks
  Interventions: Biological: Fabrazyme (agalsidase beta)

INTERVENTIONS:
Biological: Fabrazyme (agalsidase beta) — 1 mg/kg every 2 weeks
  Other Names: r-hαGAL

SUMMARY:
People with Fabry disease have an alteration in their genetic material (DNA) which causes a deficiency of the a-galactosidase A enzyme. This enzyme helps to break down and remove certain types of fatty substances called "glycolipids". These glycolipids are normally present within the body in most cells. In people with Fabry disease, glycolipids build up in various tissues such as the liver, kidney, skin, and blood vessels because a-galactosidase A is not present, or is present in small quantities. The build up of glycolipid levels (also referred to as "globotriaosylceramide" or "GL-3") in these tissues is thought to cause the clinical symptoms that are common to Fabry disease. Symptoms commonly appear during childhood with pain in the hands and feet. This study explored the safety, efficacy and pharmacokinetics of Fabrazyme in pediatric patients aged between 7 and 15 years.

ELIGIBILITY:
Inclusion criteria:

* Patient or legal guardian must provide written informed consent
* Patients must have a clinical diagnosis of Fabry disease and active Fabry disease (clinical signs and symptoms)
* Patients must be at least 7 years of age but no older than 15 years of age at time of enrollment
* Patients must be Tanner Stage ≤ III
* Female patients must have a negative pregnancy test prior to each infusion and use a medically accepted form of contraception throughout the study

Exclusion Criteria:

* Patient has a clinically significant organic disease (with the exception of symptoms relating to Fabry disease) that in the opinion of the investigator would preclude participation in the trial
* Patient has participated in a study employing investigational drug within 30 days of the start of this study
* Patient has received prior treatment with enzyme replacement therapy
* Patient is unable to comply with the clinical protocol

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2002-10; Primary Completion 2005-05 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (7):
- University of Arizona, Tucson, Arizona, United States
- France (3):
  - Hopital Edouard Herriot, Lyon
  - Hopital de la Timone Enfants, Marseille
  - Hopital Europeen Georges Pompidou, Paris
- Instytut Pomnik Centrum Zdrowia Dziecka, Warsaw, Poland
- United Kingdom (2):
  - Royal Manchester Children's Hospital, Pendlebury, Manchester
  - Great Ormond Street Hospital for Sick Children, London

REFERENCES:
- [Derived] Wraith JE, Tylki-Szymanska A, Guffon N, Lien YH, Tsimaratos M, Vellodi A, Germain DP. Safety and efficacy of enzyme replacement therapy with agalsidase beta: an international, open-label study in pediatric patients with Fabry disease. J Pediatr. 2008 Apr;152(4):563-70, 570.e1. doi: 10.1016/j.jpeds.2007.09.007. Epub 2007 Dec 3. PMID 18346516

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Fabrazyme
Started | 16
Completed | 15
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Fabrazyme
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.1 (2.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Globotriaosylceramide (GL-3) Clearance in Capillary Endothelium in the Skin
Description: Skin biopsies were taken at Baseline, Week 24 and Week 48 and analyzed for cellular GL-3 accumulation (inclusions) by light microscopy. Each biopsy was evaluated by pathologists for the total number of vessels with GL-3 accumulation on an inclusion severity score of 0 (none/trace), 1 (mild), 2 (moderate), and 3 (severe).
Time Frame: Baseline, Week 24 and Week 48
Population: Intent to Treat (ITT) population - male patients only. 14 patients had skin biopsies performed at Baseline and Week 24 but only 5 patients had skin biopsies performed at Week 48.
Measure: Number; unit: patients
Arm/Group | Fabrazyme
Number analyzed (Participants) | 14
patients
  None/Trace (0) Score at Baseline | 2
  None/Trace (0) Score at Week 24 | 14
  None/Trace (0) Score at Week 48 | 5
  Mild (1) Score at Baseline | 0
  Mild (1) Score at Week 24 | 0
  Mild (1) Score at Week 48 | 0
  Moderate (2) Score at Baseline | 11
  Moderate (2) Score at Week 24 | 0
  Moderate (2) Score at Week 48 | 0
  Severe (3) Score at Baseline | 1
  Severe (3) Score at Week 24 | 0
  Severe (3) Score at Week 48 | 0

2. Secondary Outcome: Plasma GL-3
Description: Plasma GL-3 values at Baseline, Week 24, and Week 48. Normal plasma GL-3 level is ≤ 7.03 µg/mL.
Time Frame: Baseline, Week 24 and Week 48
Population: ITT population. 16 male patients had plasma GL-3 values at Baseline and Week 24, while 15 male patients had plasma GL-3 values at Week 48. 2 female patients had plasma GL-3 values at Baseline, Week 24 and Week 48.
Measure: Mean (Standard Deviation); unit: µg/mL
Arm/Group | Fabrazyme
Number analyzed (Participants) | 16
µg/mL
  Male Patients at Baseline | 15.4 (4.10)
  Female Patients at Baseline | 4.9 (0.64)
  Overall at Baseline | 14.1 (5.25)
  Males at Week 24 | 5.5 (0.95)
  Females at Week 24 | 3.6 (0.57)
  Overall at Week 24 | 5.2 (1.10)
  Males at Week 48 | 5.0 (1.00)
  Females at Week 48 | 4.4 (1.27)
  Overall at Week 48 | 4.9 (1.01)

ADVERSE EVENTS:
Description: In the event a single participant has experienced both a serious and a non-serious form of the same adverse event term, the individual has been included in the numerator ("number of affected participants") of both adverse event tables.
Arm/Group | Fabrazyme
Serious Adverse Events (participants affected / at risk) | 1/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme (N=16)
Anaphylactic shock (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fabrazyme (N=16)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eye oedema (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 2
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 7
Abdominal pain upper (Gastrointestinal disorders) | 4
Chapped lips (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 5
Dyspepsia (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 9
Toothache (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 9
Asthenia (General disorders) | 2
Catheter site pain (General disorders) | 1
Chest pain (General disorders) | 2
Chills (General disorders) | 3
Fatigue (General disorders) | 1
Feeling cold (General disorders) | 2
Feeling hot (General disorders) | 2
Hyperthermia (General disorders) | 1
Injection site pain (General disorders) | 1
Malaise (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 7
Seasonal allergy (Immune system disorders) | 1
Gastroenteritis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 4
Pharyngitis (Infections and infestations) | 4
Tonsillitis (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Concussion (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Joint injury (Injury, poisoning and procedural complications) | 1
Joint sprain (Injury, poisoning and procedural complications) | 2
Post-traumatic pain (Injury, poisoning and procedural complications) | 1
Procedural complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Testicular injury (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Albumin urine present (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Body temperature increased (Investigations) | 3
Creatinine renal clearance decreased (Investigations) | 1
Heart rate increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 3
Cognitive disorder (Nervous system disorders) | 1
Coordination abnormal (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Dyspraxia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 10
Hyperreflexia (Nervous system disorders) | 1
Lethargy (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 6
Tremor (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Microalbuminuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1
Angiokeratoma (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Urticaria localised (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1
Pallor (Vascular disorders) | 1
Poor peripheral circulation (Vascular disorders) | 1
Vasoconstriction (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The trial was not powered to demonstrate clinical benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In multi-site studies, PI can publish after Genzyme publishes or 18 months after study completion. PI gives Genzyme a draft 60 days before publication. Genzyme can ask that confidential information be removed, and can defer publication another 60 days upon notifying PI that it will file a patent application on inventions contained in the draft.